CLINICAL TRIAL: NCT01403025
Title: A Multi-centre, Open Label, Observational, Non-interventional Study to Evaluate the Safety and Effectiveness of Victoza® in Subjects With Type 2 Diabetes Mellitus
Brief Title: Evaluating the Safety and Effectiveness of Liraglutide in Subjects With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3772; U1111-1120-7575 (Other: WHO); JapicCTI-111559 (Registry Identifier: JAPIC)
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Once daily at a fixed timing, and subcutaneously (under the skin) in the abdomen, in the thigh or in the upper arm

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to assess the incidence rate and type of SADRs (serious adverse drug reactions).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus, including newly-diagnosed subjects, who require treatment with liraglutide

Exclusion Criteria:

* Subjects who are or have previously been on liraglutide
* Subjects who have previously been enrolled in the study
* Subjects with a hypersensitivity to liraglutide or to any of the excipients
* Subjects who are pregnant, breast feeding or have the intention of becoming pregnant within the study periods
* Subjects with cancer (except basal cell skin cancer or squamous cell skin cancer) or any clinically significant disorder, except for conditions associated with type 2 diabetes mellitus history which in the physicians' opinion could interfere with the results of the trial
* Known or suspected abuse of alcohol or narcotics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with type 2 diabetes mellitus, including newly-diagnosed subjects, who are considered to need treatment with liraglutide (Victoza®)
Sampling Method: Non-Probability Sample
Enrollment: 4121 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2015-12-28 (Actual); Study Completion 2015-12-28 (Actual)

PRIMARY OUTCOMES:
The incidence of SADRs (Serious Adverse Drug Reactions) | After 36 months

SECONDARY OUTCOMES:
The incidence rate and type of SAEs (Serious Adverse Events) | At month 1, 3, 6, 12, 24 and 36
The incidence rate and type of ADRs (Adverse Drug Reactions) | At month 1, 3, 6, 12, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com